CLINICAL TRIAL: NCT06577831
Title: Dynamic Monitoring and Characterization of Pelvic by 3D Ultrafast MRI
Acronym: DYNPELVIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RCAPHM20_0016
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Pelvic Deformity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient (Experimental): Patients requiring dynamic MRI for the diagnosis of pelvic static disorders
  Interventions: Diagnostic Test: dynamic MRI
- control (Active Comparator): Healthy volunteers for a dynamic MRI
  Interventions: Diagnostic Test: dynamic MRI

INTERVENTIONS:
Diagnostic Test: dynamic MRI — * MRI sequences will be performed for patients and healthy volunteers i
  * Vaginal and rectal tagging will be performed using a water-based ultrasound gel.
  * The gel will be inserted by an authorized person (nurse or doctor) using a syringe with a conical tip and, optionally, a probe.
  * MRI sequences.
  * Data analysis and interpretation.

SUMMARY:
Pelvic floor disorders affect a large population of women and are responsible for a significant impairment in their quality of life, but the pathophysiology of these disorders is still poorly understood.

The project proposes to define new ultra-fast 3D MRI sequences to capture the movements of the main pelvic organs. Visualization of 3D volumes is of great importance to clinicians, but data size hinders clinical use.

This study is the first to propose a dynamic 3D representation of pelvic organs, together with quantitative estimates of the deformations undergone.

The method is based on four steps: dynamic acquisition, organ segmentation, temporal reconstruction, quantification and visualization of deformations.

The D3-Pelvis project responds to the challenge of "technologies for health" with dynamic 3D MRI acquisition and 3D modeling, offering prospects for diagnostic aids and simulators.

ELIGIBILITY:
Inclusion Criteria:

* Adult women, +/- of childbearing age, with or without effective contraception.
* Informed consent signed prior to any procedure described in the study.

Exclusion Criteria:

* Contraindication to MRI,
* Impossibility of performing the examination during thrust,
* Minor patients
* Pregnant or breast-feeding women,
* Women of legal age under guardianship
* Persons staying in a health or social institution,
* People in emergency situations,
* Persons not covered by a social security scheme,
* Persons deprived of their liberty.
* Specifically, women with IUDs will be excluded if they cannot remove them before the examination.
* For healthy volunteers: history of colorectal surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Develop new three-dimensional analysis tools combining high spatial resolution static MRI with ultra-fast dynamic MRI. | 0 month
  a metric for displacement of the anchor points of the targeted pelvic organs will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hopitaux de Marseille _ Hopital de la Timone, Marseille, France, France

IPD SHARING:
Plan to Share IPD: No